CLINICAL TRIAL: NCT03243422
Title: Aging and Cognitive Health Evaluation in Elders (ACHIEVE) Randomized Trial
Brief Title: Aging and Cognitive Health Evaluation in Elders (ACHIEVE)
Acronym: ACHIEVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: University of North Carolina (Other); University of South Florida (Other); University of Pittsburgh (Other); University of Mississippi Medical Center (Other); Wake Forest University (Other); University of Minnesota (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00008129; R01AG055426 (NIH)
Record Dates: First submitted 2017-07-27; First posted 2017-08-09 (Actual); Results first posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Aging; Cognitive Decline
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Successful aging health education intervention (Active Comparator): Individual sessions on healthy aging topics
  Interventions: Other: Successful aging health education intervention
- Hearing intervention (Active Comparator): Best practices hearing rehabilitative treatment
  Interventions: Other: Hearing intervention

INTERVENTIONS:
Other: Successful aging health education intervention — The Successful Aging intervention will follow the protocol and materials developed for the 10 Keys™ to Healthy Aging program by the Center for Aging and Population Health Prevention Research Center at the University of Pittsburgh. This interactive, dynamic program informs older adults about risk factors for diseases. Participants will meet individually with a health educator certified to administer the program every 2-3 weeks for a total of 4 visits over approximately 8-10 weeks, and the session content will focus on a "Key". Each session will also include a 5-10 minute active upper body extremity stretching program as used in the Lifestyle Interventions and Independence for Elders (LIFE) study. Participants will return for booster sessions semi-annually beginning at 6 months post-randomization.
  Arms: Successful aging health education intervention
Other: Hearing intervention — The hearing intervention consists of fitting with hearing aids and other hearing assistive technologies plus four 1-hour comprehensive, individualized hearing rehabilitation sessions spaced over the 2-3 months post-randomization designed to provide all of the active components of the intervention. Hearing aids are instructed to be worn on a daily basis for study duration. Audiologic outcomes (e.g., hearing aid data logging, real ear measures, speech in noise, etc.) to verify the best-practices hearing intervention are gathered during study intervention visits and semi-annually beginning at 6 months post-randomization.
  Arms: Hearing intervention

SUMMARY:
The ACHIEVE study will be a randomized controlled trial nested within the infrastructure of the Atherosclerosis Risk in Communities (ARIC) study. We plan to enroll 850 70-84 year-old cognitively normal older adults with hearing loss, who will be randomized 1:1 to the hearing intervention (hearing needs assessment, fitting of hearing devices, education/counseling) or successful aging health education intervention (individual sessions with a health educator covering healthy aging topics). Post-baseline, participants will be followed semi-annually for 3 years.

DETAILED DESCRIPTION:
The ACHIEVE study will be a randomized controlled trial nested within the infrastructure of the Atherosclerosis Risk in Communities (ARIC) study. We plan to enroll 850 70-84 year-old cognitively normal older adults with hearing loss, who will be randomized 1:1 to the hearing intervention (hearing needs assessment, fitting of hearing devices, education/counseling) or successful aging health education intervention (individual sessions with a health educator covering healthy aging topics). Post-baseline, participants will be followed semi-annually for 3 years.

Outcomes will include assessments of cognition, social functioning, physical functioning, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age 70-84 years. Individuals aged 70-84 at the time of randomization are eligible for participation. This age range will allow recruitment of participants who are at risk for cognitive decline but who may also be expected to survive for the duration of the trial. This age range is estimated to allow for potential participation of 61% of participants currently enrolled in the ARIC study.
* Community-dwelling.
* Fluent English-speaker.
* Residency. Participants must plan to reside in the local area for the study duration.
* Audiometric hearing impairment. Participants must have adult-onset hearing impairment with a four-frequency pure tone average (0.5, 1, 2, 4 kHz) in the better-hearing ear of ≥ 30 decibels (dB) and <70 dB. This level of hearing impairment is the level at which individuals would be most likely to benefit from the use of conventional amplification devices such as hearing aids.
* Word Recognition in Quiet score ≥60% in the better ear. A word recognition in quiet score <60% suggests hearing impairment that is too severe to benefit from conventional amplification devices such as hearing aids.
* Mini-Mental State Exam (MMSE) score ≥ 23 for individuals with high-school degree or less; Mini-Mental State Exam (MMSE) score ≥ 25 for individuals with some college or more; Participants must be at risk for cognitive decline in the range quantified well by neurocognitive testing, and so must be free from more substantial cognitive impairment at baseline.
* Willingness to participate be randomized and adhere to the protocol. Participants must be willing and able to consent to participate in the study, be willing to be randomized to either the Hearing intervention or to the Successful Aging intervention, and be willing to commit to adhere to the study protocol for the duration of the trial (3 years of a randomly assigned intervention).

Exclusion Criteria:

* Self-reported disability in ≥ 2 or more Activities of Daily Living (ADL).
* Any self-reported hearing aid use in the past year. Trial participants will be randomized to hearing intervention or successful aging intervention and, therefore, participants cannot be receiving treatment for their hearing loss already.
* ARIC participants only: Diagnosis of adjudicated dementia based on a previous ARIC visit or participant required a proxy to assist with completing informed consent and responding to questions at ARIC Visit 6 or 7.
* Vision impairment (worse than 20/63 on MNREAD Acuity Chart). Participants who cannot see (with correction) well enough to complete the neurocognitive assessment are excluded.
* Medical contraindication to use of hearing aids (e.g., draining ear). Because hearing aids will be the primary device used in the hearing intervention, participants with medical contraindications to hearing aid use are excluded.
* Permanent conductive hearing impairment as determined by a difference in air audiometry and bone audiometry ("air-bone gap") greater than 15 dB in 2 or more contiguous frequencies in both ears. Because the impact of a conductive (versus a sensorineural) hearing loss on cognitive functioning may potentially differ and programming for hearing aids differs for conductive hearing loss, participants with permanent conductive hearing loss are excluded from the trial. Participants with an air-bone gap due to fluid in the ears or other resolvable medical issue may be enrolled in the trial following successful medical resolution of the cause of the air-bone gap.
* Unwilling to wear hearing aids on a regular (i.e., daily or near daily) basis.

Ages: 70 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 977 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank R Lin, MD, PhD, Principal Investigator — Johns Hopkins University; Josef Coresh, Principal Investigator — Johns Hopkins University
Locations (4):
- United States (4):
  - Johns Hopkins Comstock Center for Public Health Research, Hagerstown, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Wake Forest University, Winston-Salem, North Carolina

REFERENCES:
- [Derived] Goman AM, Tan N, Pike JR, Bessen SY, Chen ZS, Huang AR, Arnold ML, Burgard S, Chisolm TH, Couper D, Deal JA, Glynn NW, Gmelin T, Gravens-Mueller L, Hayden KM, Martinez-Amezcua P, Mitchell CM, Pankow JS, Reed NS, Sanchez VA, Schrack JA, Sullivan KJ, Coresh J, Lin FR; ACHIEVE Collaborative Research Group. Effects of hearing intervention on falls in older adults: findings from a secondary analysis of the ACHIEVE randomised controlled trial. Lancet Public Health. 2025 Jun;10(6):e492-e502. doi: 10.1016/S2468-2667(25)00088-X. PMID 40441816
- [Derived] Pike JR, Huang AR, Reed NS, Arnold M, Chisolm T, Couper D, Deal JA, Glynn NW, Goman AM, Hayden KM, Mitchell CM, Pankow JS, Sanchez V, Sullivan KJ, Tan NS, Coresh J, Lin FR; ACHIEVE Collaborative Research Group. Cognitive benefits of hearing intervention vary by risk of cognitive decline: A secondary analysis of the ACHIEVE trial. Alzheimers Dement. 2025 May;21(5):e70156. doi: 10.1002/alz.70156. PMID 40369891
- [Derived] Reed NS, Chen J, Huang AR, Pike JR, Arnold M, Burgard S, Chen Z, Chisolm T, Couper D, Cudjoe TKM, Deal JA, Goman AM, Glynn NW, Gmelin T, Gravens-Mueller L, Hayden KM, Mitchell CM, Mosley T, Oh ES, Pankow JS, Sanchez VA, Schrack JA, Coresh J, Lin FR; ACHIEVE Collaborative Research Group. Hearing Intervention, Social Isolation, and Loneliness: A Secondary Analysis of the ACHIEVE Randomized Clinical Trial. JAMA Intern Med. 2025 Jul 1;185(7):797-806. doi: 10.1001/jamainternmed.2025.1140. PMID 40354063
- [Derived] Huang AR, Morales EG, Arnold ML, Burgard S, Couper D, Deal JA, Glynn NW, Gmelin T, Goman AM, Gravens-Mueller L, Hayden KM, Mitchell CM, Pankow JS, Pike JR, Reed NS, Sanchez VA, Schrack JA, Sullivan KJ, Coresh J, Lin FR, Chisolm TH; ACHIEVE Collaborative Research Group. A Hearing Intervention and Health-Related Quality of Life in Older Adults: A Secondary Analysis of the ACHIEVE Randomized Clinical Trial. JAMA Netw Open. 2024 Nov 4;7(11):e2446591. doi: 10.1001/jamanetworkopen.2024.46591. PMID 39570588
- [Derived] Lin FR, Pike JR, Albert MS, Arnold M, Burgard S, Chisolm T, Couper D, Deal JA, Goman AM, Glynn NW, Gmelin T, Gravens-Mueller L, Hayden KM, Huang AR, Knopman D, Mitchell CM, Mosley T, Pankow JS, Reed NS, Sanchez V, Schrack JA, Windham BG, Coresh J; ACHIEVE Collaborative Research Group. Hearing intervention versus health education control to reduce cognitive decline in older adults with hearing loss in the USA (ACHIEVE): a multicentre, randomised controlled trial. Lancet. 2023 Sep 2;402(10404):786-797. doi: 10.1016/S0140-6736(23)01406-X. Epub 2023 Jul 18. PMID 37478886
- [Derived] Sanchez VA, Arnold ML, Reed NS, Oree PH, Matthews CR, Clock Eddins A, Lin FR, Chisolm TH. The Hearing Intervention for the Aging and Cognitive Health Evaluation in Elders Randomized Control Trial: Manualization and Feasibility Study. Ear Hear. 2020 Sep/Oct;41(5):1333-1348. doi: 10.1097/AUD.0000000000000858. PMID 32251012
- [Derived] Deal JA, Goman AM, Albert MS, Arnold ML, Burgard S, Chisolm T, Couper D, Glynn NW, Gmelin T, Hayden KM, Mosley T, Pankow JS, Reed N, Sanchez VA, Richey Sharrett A, Thomas SD, Coresh J, Lin FR. Hearing treatment for reducing cognitive decline: Design and methods of the Aging and Cognitive Health Evaluation in Elders randomized controlled trial. Alzheimers Dement (N Y). 2018 Oct 5;4:499-507. doi: 10.1016/j.trci.2018.08.007. eCollection 2018. PMID 30364572

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants were randomized using 1:1 permuted block randomization, stratified by severity of hearing loss (PTA <40 dB or ≥ 40 dB), recruitment source (ARIC or de novo), and field site, to either hearing intervention (HI) or a successful aging (SA) health education control intervention from January 2018 to October 2019. Eligible participants who were spouses/partners were randomized as a unit, stratified by recruitment source and field site.
Period: Overall Study
Arm/Group | Successful Aging Health Education Intervention | Hearing Intervention
Started | 487 | 490
Completed | 436 | 440
Not Completed | 51 | 50
Not completed — Death | 20 | 21
Not completed — Lost to Follow-up | 9 | 21
Not completed — Withdrawal by Subject | 22 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Successful Aging Health Education Intervention | Hearing Intervention | Total
Number analyzed (Participants) | 487 | 490 | 977
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 487 | 490 | 977
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Overall there were 977 participants enrolled, 238 were from ARIC and 739 were from De Novo
  years
    Overall | 77.0 (4.0) | 76.5 (3.9) | 76.8 (4.0)
    ARIC participants: number analyzed (Participants) | 118 | 120 | 238
    ARIC participants | 78.6 (2.9) | 79.2 (2.9) | 78.9 (2.9)
    De Novo participants: number analyzed (Participants) | 369 | 370 | 739
    De Novo participants | 76.5 (4.2) | 75.7 (3.8) | 76.1 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Overall: Female | 259 | 264 | 523
  Overall: Male | 228 | 226 | 454
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 59 | 53 | 112
  White | 424 | 434 | 858
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 487 | 490 | 977
Recruitment Source [Count of Participants; unit: Participants]
  ARIC | 118 | 120 | 238
  De Novo | 369 | 370 | 739
Field Sites [Count of Participants; unit: Participants]
  Forsyth County, NC | 119 | 117 | 236
  Jackson, MI | 123 | 120 | 243
  Minneapolis, Mn | 116 | 120 | 236
  Washington County, MD | 129 | 133 | 262
4-Frequency pure tone average dB [Mean (Standard Deviation); unit: dB] | 39.3 (6.7) | 39.5 (7.1) | 39.4 (6.9)
Education (highest level obtained) [Count of Participants; unit: Participants]
  Less than high school | 18 | 19 | 37
  High school, GED, or vocational school | 212 | 206 | 418
  College, graduate, or professional school | 257 | 264 | 521
  Missing | 0 | 1 | 1
APOE E4 gene [Count of Participants; unit: Participants]
  APOE gene present | 114 | 110 | 224
  APOE gene not present | 345 | 339 | 684
  Missing | 28 | 41 | 69

OUTCOME MEASURES:

1. Primary Outcome: Change in Global Cognitive Function
Description: Mean change in global cognitive function in standard deviations from baseline to year 3 estimated from a linear mixed-effects model. Global cognitive function was defined as a factor score derived from the completion of a neurocognitive testing battery. The ACHIEVE study administers a neurocognitive testing battery annually, which includes the following cognitive tests: Delayed Word Recall, Consortium to Establish a Registry for Alzheimer's Disease (CERAD) Word List, Incidental Learning, Logical Memory I and II, Word Fluency, Animal Naming, Boston Naming, Trail Making Test A and B, Digit Span Backwards, and Digit Symbol Substitution. Factor analytic methods use all items from all tests in the battery to generate a single score of global cognitive function. The global cognitive function factor score has a minimum of -5 and a maximum of 4. Lower scores denote worse cognitive function.
Time Frame: 3 years
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Successful Aging Health Education Intervention | Hearing Intervention
Number analyzed (Participants) | 487 | 490
score on a scale | -0.202 [-0.258 to -0.145] | -0.200 [-0.256 to -0.144]
Statistical Analysis 1: Comparison: Successful Aging Health Education Intervention; Test type: Superiority; p = 0.96, Mixed Models Analysis; Three-level linear mixed effects model with an unstructured covariance matrix from the baseline and the year 3 in-person neurocognitive assessment; change in Standard Deviation = 0.002, 95% CI 2-sided [-0.077 to 0.081]

2. Secondary Outcome: Change in Cognition Memory Domain
Description: Mean change in cognition memory domain in standard deviations from baseline to year 3 estimated from a linear mixed-effects model. The cognition memory domain was defined as a factor score derived from the completion of a neurocognitive testing battery. The cognitive tests for the memory domain include Delayed Word Recall, CERAD Word List, Incidental Learning, and Logical Memory I and II. These tests have an underlying commonality or factor, that is unable to be directly measured, and factor analytic methods use items from the tests noted to generate a single overall memory score. The cognition memory domain factor score has a minimum of -5 and a maximum of 4. Lower scores denote worse cognitive function.
Time Frame: 3 years
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Successful Aging Health Education Intervention | Hearing Intervention
Number analyzed (Participants) | 487 | 490
score on a scale | -0.054 [-0.128 to 0.020] | 0.025 [-0.053 to 0.103]
Statistical Analysis 1: Comparison: Successful Aging Health Education Intervention vs Hearing Intervention; Test type: Superiority; p = 0.15, Mixed Models Analysis — Secondary outcomes were evaluated with Hochberg modification to the Bonferroni adjustment estimates are considered statistically significant if the largest p-value is <0·05; Slope = 0.079, 95% CI 2-sided [-0.029 to 0.187]

3. Secondary Outcome: Change in Cognition Executive Function Domain
Description: Mean change in cognitive executive function in standard deviations from baseline to year 3 estimated from a linear mixed-effects model. The executive function domain was defined as a factor score derived from the completion of a neurocognitive testing battery. The cognitive tests for the executive function domain include Trail Making Test A and B and Digit Symbol Substitution. These tests have an underlying commonality or factor, that is unable to be directly measured, and factor analytic methods use items from the tests noted to generate a single overall executive function score. The executive function cognitive factor score has a minimum of -5 and a maximum of 4. Lower scores denote worse cognitive function.
Time Frame: 3 years
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Successful Aging Health Education Intervention | Hearing Intervention
Number analyzed (Participants) | 487 | 490
score on a scale | -0.248 [-0.315 to -0.181] | -0.268 [-0.339 to -0.197]
Statistical Analysis 1: Comparison: Successful Aging Health Education Intervention vs Hearing Intervention; Test type: Superiority; p = 0.69, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Slope = -0.020, 95% CI 2-sided [-0.118 to 0.078]

4. Secondary Outcome: Change in Cognition Language Domain
Description: Mean change in cognition language domain in standard deviations from baseline to year 3 estimated from a linear mixed-effects model. The cognition language domain as defined as a factor score derived from the completion of a neurocognitive testing battery. The cognitive tests for the language domain include Word Fluency, Animal Naming, and Boston Naming. These tests have an underlying commonality or factor, that is unable to be directly measured, and factor analytic methods use items from the tests noted to generate a single overall language score. The cognition language domain factor score has a minimum of -5 and a maximum of 4. Lower scores denote worse cognitive function.
Time Frame: 3 years
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Successful Aging Health Education Intervention | Hearing Intervention
Number analyzed (Participants) | 487 | 490
score on a scale | -0.155 [-0.214 to -0.096] | -0.138 [-0.199 to -0.077]
Statistical Analysis 1: Comparison: Successful Aging Health Education Intervention vs Hearing Intervention; Test type: Superiority; p = 0.70, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Slope = 0.017, 95% CI 2-sided [-0.070 to 0.104]

5. Secondary Outcome: Number of Participants Who Developed Cognitive Impairment
Description: Incident cognitive impairment with the outcome defined as the first instance of (1) adjudicated diagnosis of dementia or mild cognitive impairment (MCI), (2) 3-point drop in the 30-item Mini-Mental State Exam (MMSE) administered in-person, or (3) a 3-point drop in a factor score derived from the 10-item MMSE orientation subscale and 11-item Blessed scale administered over the telephone and rescaled to be equivalent to the 30-item MMSE. The numbers below in the outcome measure data table represent the number of cases (participants) who developed cognitive impairment, within 3 years.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Successful Aging Health Education Intervention | Hearing Intervention
Number analyzed (Participants) | 487 | 490
Participants | 49 | 45
Statistical Analysis 1: Comparison: Successful Aging Health Education Intervention vs Hearing Intervention; Test type: Superiority; p = 0.59, Regression, Cox — [p-value comment as in outcome 2, analysis 1]; Discrete-time interval model; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.61 to 1.33]

6. Other Pre Specified Outcome: 3-year Global Cognitive Change Restricted to ARIC Participants
Description: Mean change in global cognitive function in standard deviations from baseline to year 3 estimated from a linear mixed-effects model. Global cognitive function was defined as a factor score derived from the completion of a neurocognitive testing battery. The ACHIEVE study administers a neurocognitive testing battery annually, which includes the following cognitive tests: Delayed Word Recall, Consortium to Establish a Registry for Alzheimer's Disease (CERAD) Word List, Incidental Learning, Logical Memory I and II, Word Fluency, Animal Naming, Boston Naming, Trail Making Test A and B, Digit Span Backwards, and Digit Symbol Substitution. Factor analytic methods use all items from all tests in the battery to generate a single score of global cognitive function. The global cognitive function factor score has a minimum of -5 and a maximum of 4. Lower scores denote worse cognitive function. Stratified by recruitment type ARIC vs De Novo.
Time Frame: 3 year
Population: ARIC participants participating in ACHIEVE were randomized to either hearing intervention or successful aging health education intervention.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- ARIC Only Successful Aging Health Education Intervention: Individual sessions on healthy aging topics
  Successful aging health education intervention: The Successful Aging intervention will follow the protocol and materials developed for the 10 Keys™ to Healthy Aging program by the Center for Aging and Population Health Prevention Research Center at the University of Pittsburgh. This interactive, dynamic program informs older adults about risk factors for diseases. Participants will meet individually with a health educator certified to administer the program every 2-3 weeks for a total of 4 visits over approximately 8-10 weeks, and the session content will focus on a "Key". Each session will also include a 5-10 minute active upper body extremity stretching program as used in the Lifestyle Interventions and Independence for Elders (LIFE) study. Participants will return for booster sessions semi-annually beginning at 6 months post-randomization.
- ARIC Only Hearing Intervention: Best practices hearing rehabilitative treatment
  Hearing intervention: The hearing intervention consists of fitting with hearing aids and other hearing assistive technologies plus four 1-hour comprehensive, individualized hearing rehabilitation sessions spaced over the 2-3 months post-randomization designed to provide all of the active components of the intervention. Hearing aids are instructed to be worn on a daily basis for study duration. Audiologic outcomes (e.g., hearing aid data logging, real ear measures, speech in noise, etc.) to verify the best-practices hearing intervention are gathered during study intervention visits and semi-annually beginning at 6 months post-randomization.
Arm/Group | ARIC Only Successful Aging Health Education Intervention | ARIC Only Hearing Intervention
Number analyzed (Participants) | 118 | 120
score on a scale | -0.402 [-0.536 to -0.267] | -0.211 [-0.349 to -0.073]
Statistical Analysis 1: Comparison: ARIC Only Successful Aging Health Education Intervention vs ARIC Only Hearing Intervention; Analysis was restricted to ARIC participants who were enrolled in ACHIEVE; Test type: Superiority; p = 0.027, Mixed Models Analysis; Slope = 0.191, 95% CI 2-sided [0.022 to 0.360]

7. Other Pre Specified Outcome: 3-year Global Cognitive Change Restricted to De Novo Participants
Description: as for outcome 6
Time Frame: 3 year
Population: De Novo participants participating in ACHIEVE were randomized to either hearing intervention or successful aging health education intervention.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- De Novo Only Successful Aging Health Education Intervention: Individual sessions on healthy aging topics
  Successful aging health education intervention: The Successful Aging intervention will follow the protocol and materials developed for the 10 Keys™ to Healthy Aging program by the Center for Aging and Population Health Prevention Research Center at the University of Pittsburgh. This interactive, dynamic program informs older adults about risk factors for diseases. Participants will meet individually with a health educator certified to administer the program every 2-3 weeks for a total of 4 visits over approximately 8-10 weeks, and the session content will focus on a "Key". Each session will also include a 5-10 minute active upper body extremity stretching program as used in the Lifestyle Interventions and Independence for Elders (LIFE) study. Participants will return for booster sessions semi-annually beginning at 6 months post-randomization.
- De Novo Only Hearing Intervention: Best practices hearing rehabilitative treatment
  Hearing intervention: The hearing intervention consists of fitting with hearing aids and other hearing assistive technologies plus four 1-hour comprehensive, individualized hearing rehabilitation sessions spaced over the 2-3 months post-randomization designed to provide all of the active components of the intervention. Hearing aids are instructed to be worn on a daily basis for study duration. Audiologic outcomes (e.g., hearing aid data logging, real ear measures, speech in noise, etc.) to verify the best-practices hearing intervention are gathered during study intervention visits and semi-annually beginning at 6 months post-randomization.
Arm/Group | De Novo Only Successful Aging Health Education Intervention | De Novo Only Hearing Intervention
Number analyzed (Participants) | 369 | 370
score on a scale | -0.151 [-0.215 to -0.087] | -0.213 [-0.277 to -0.148]
Statistical Analysis 1: Comparison: De Novo Only Successful Aging Health Education Intervention vs De Novo Only Hearing Intervention; Test type: Superiority; p = 0.18, Mixed Models Analysis; Slope = -0.061, 95% CI 2-sided [-0.151 to 0.028]

8. Other Pre Specified Outcome: Social Engagement
Description: Change from baseline to year 3 in social engagement, as assessed by the Cohen's Social Network Index (SNI) questionnaire, which asks about the number of people the participant has regular contact with (at least once every 2 weeks) within each of 12 different possible settings/types of contacts (e.g., relatives, church members, neighbors, etc.). Social engagement is quantified by evaluating the total number of people in the social network across all 12 settings/roles.
Time Frame: 3 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Loneliness
Description: Change from baseline to year 3 in loneliness, as assessed using the University of California Los Angeles (UCLA) Loneliness Scale questionnaire. The UCLA Loneliness Scale is interviewer administered and consists of 20 items that participants rate using a 4-point Likert scale; 9 positively worded items are reverse-coded, and the average scores range from 1 to 4, with higher score indicating greater expression of loneliness.
Time Frame: 3 years
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Physical Function: Lower Extremity Function
Description: Change from baseline to year 3 in lower extremity function, as assessed using the Short Physical Performance Battery (SPPB), which includes timed tests for usual gait speed, balance, and the ability to rise from a chair. Each of the 3 tests is scored from 0 to 4, with higher scores reflecting better lower extremity physical performance, and the total SPPB score is calculated as the sum of the 3 tests, with a range of 0 to 12, with higher scores reflecting better physical performance.
Time Frame: 3 years
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Physical Function: Grip Strength
Description: Change from baseline to year 3 in grip strength (kilograms of force) measured by a hand-held dynamometer, based on the best of two trials with the participant's preferred or best hand.
Time Frame: 3 years
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Physical Function: Physical Activity
Description: Change from baseline to year 3 in physical activity measured by accelerometry. Participants will use a wrist-worn device that is worn continuously for 7 days after baseline, and 7 days after each annual follow up. This measures the intensity, duration, and frequency of physical activity.
Time Frame: 3 years
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Self-reported Physical Ability
Description: Change from baseline to year 3 measured using the falls and mobility questionnaire which records living circumstances, self-reported physical ability, fatigue, and falls.
Time Frame: 3 years
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Self-reported Physical Activity
Description: Change from baseline to year 3 in self-reported physical activity measured using the Baecke Physical Activity Questionnaire, which includes questions about frequency of exercise/sports and leisure activities to generate composite scores of sports during leisure time (continuous measure between 1 and 5) and leisure time excluding sports (continuous measure between 1 and 5).
Time Frame: 3 years
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Depressive Symptoms
Description: Change from baseline to year 3 in depressive symptoms, as assessed by the Center for Epidemiological Studies Depression Scale (CES-D). The CES-D is an interviewer-administered scale that consists of 12 items which participants rate using a 3-point Likert scale; 2 positively worded items are reverse-coded. The first 11 items are summed to create a total score ranging from 0 to 22, with higher scores indicating greater expression of depression. The 12th item is a rating of hopelessness that is not included in the total score.
Time Frame: 3 years
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Hearing Handicap
Description: Change from baseline to year 3 measured on the Hearing Handicap for the Elderly Screening Version (HHIE-S) questionnaire, which is a 10-item questionnaire developed to assess how an individual perceives the social and emotional effects of hearing loss; scores range from 0 to 40, with higher scores suggestive of greater hearing handicap
Time Frame: 3 years
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Intervention Feedback
Description: A questionnaire that gathers feedback about the study intervention that participants are receiving. Participants rate how strongly they agree or disagree with a series of statements about the ACHIEVE study intervention they received.
Time Frame: Gathered at 6 months post-baseline and 36 months post-baseline
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Physical Health
Description: Change from baseline to year 3 as assessed using the RAND-36, which is an interviewer-administered scale measuring a person's perceptions of their health and health-related quality of life; the physical component score is an algorithmically derived score with a normative mean of 50 and standard deviation of 10 (range 0 to 100), where higher scores indicate better physical health.
Time Frame: 3 years
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Mental Health
Description: Change from baseline to year 3 as assessed using the RAND-36, which is an interviewer-administered scale measuring a person's perceptions of their health and health-related quality of life; the mental component score is an algorithmically derived score with a normative mean of 50 and standard deviation of 10 (range 0 to 100), where higher scores indicate better mental health.
Time Frame: 3 years
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Hospitalizations
Description: Number of hospitalizations (all cause) over the course of follow-up based on self-report
Time Frame: 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Every six months after randomization, up to 3 years.
Description: For ACHIEVE only otitis externa and cerumen impaction or ear foreign body requiring removal by a physician were considered adverse events. Death from any cause was considered a serious adverse event.
Arm/Group | Successful Aging Health Education Intervention | Hearing Intervention
All-Cause Mortality (participants affected / at risk) | 20/487 | 21/490
Serious Adverse Events (participants affected / at risk) | 0/487 | 0/490
Other Adverse Events (participants affected / at risk) | 17/487 | 41/490
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Successful Aging Health Education Intervention (N=487) | Hearing Intervention (N=490)
Otitis externa (Ear and labyrinth disorders) | 2 (2) | 9 (9) — Otitis externa (outer ear infection)
Cerumen impaction (Ear and labyrinth disorders) | 15 (15) | 28 (28) — Cerumen impaction or ear foreign body requiring removal by physician
Other (Ear and labyrinth disorders) | 0 (0) | 4 (4) — Includes left serous effusion, hearing aid dome stuck on the ear canal, fungal infection of the ear canal, and eustachian tube inflammation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-03-23): https://cdn.clinicaltrials.gov/large-docs/22/NCT03243422/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/22/NCT03243422/SAP_001.pdf